CLINICAL TRIAL: NCT00433901
Title: Managing Weight in Overweight and At-Risk Children
Brief Title: Family Connections Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Paul Estabrooks, PhD, Kaiser Permanente Institute for Health Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CO-04Esta-05
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Childhood Obesity
Keywords: obesity in children; childhood disorders; overweight children; physical activity; home environment
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

INTERVENTIONS:
Behavioral: Targeted parental instruction for positive lifestyle change with follow-up calls.

SUMMARY:
The prevalence of overweight children has increased significantly over the past 3 decades and 3 out of every 4 overweight children become obese adults. Additionally, overweight children are now at risk for developing type-2 diabetes while still in their youth. To address the issue of childhood weight management, Golan and colleagues provided a model for intervention development that targets parents as an exclusive agent of change when attempting to treat weight issues for children under 12 years of age. The Kaiser Permanente Colorado (KPCO) Weight Management Program (WMP) developed Family Connections, a condensed two-session program, based on the Golan model, for parents of children between the ages of 8-12 with a Body Mass Index (BMI) greater than the 85 percentile for age and gender. There is a need to determine if the content of Golan's model can be translated into a practical intervention to be used in usual pediatric weight management practice. The Family Connections study uses three arms to determine the effectiveness of healthy eating and active living messages.

DETAILED DESCRIPTION:
We used a 3 condition randomized controlled trial design to allow us to make comparisons across current standard care, Family Connections, and Family Connections plus telephone follow-up support.

Duration:

The study is conducted in a two year and four month period; beginning in November, 2004 and ending in February, 2007.

Description of intervention:

Workbook Control. A workbook was created from the content of the two part Family Connections classes, the current standard of care. The workbook has themes which promote increased PA and fruit & vegetable (FV) consumption in concert with decreased soda consumption (SC), and television viewing/recreational computer time (TV). Specific intervention themes included parental cognitive and behavior change, home environment change, and parental modeling of healthy behaviors.

Family Connections-current standard of care. The Family Connections classes are a two part intervention targeted toward the primary caretakers of the overweight child. The classes were held one week apart at a local Kaiser Permanente health clinic. Parents were also given a copy of the workbook to use in class and at home.

Family Connections plus Automated Telephone Follow-up. Parents assigned to this intervention arm will complete the Family Connections program and subsequently receive 10 follow-up sessions delivered via Interactive Voice Response (IVR) technology. The calls will be completed with high frequency initially and then scaled back over time. To sustain changes that are made as a result of the Family Connections program, telephone follow-up calls commenced 1 week after the second class. Calls occurred on a weekly basis for 1 month. During the 3rd and 4th month calls occurred biweekly. Finally a monthly call was provided during the 5th and 6th months of the study. The calls will include content targeted towards, increasing parental behavioral health, parenting and role modeling skills as well as providing strategies for home environmental changes to promote healthy eating and PA. In addition, a goal setting and assessment tool was provided; at the beginning of each call the primary parent would hear the goal they selected the week prior and rate their achievement. Based on the rating, the primary parent was given the option to hear tips related to the topic of their prior week's selected goal area.

Specific aims:

PRIMARY AIM 1: To determine the effectiveness (6 & 12 months after the intervention initiation) of Family Connections when compared to a standard care control group in reducing child BMI percentile rankings. Other key outcomes will be physical activity (PA) and healthy eating behaviors (i.e., ↑ fruits & vegetables; ↓Soda/sugar drinks).

PRIMARY AIM 2: To determine the effectiveness (6 & 12 months after the initiation of intervention) of adding automated telephone follow-ups using a 3 group randomized controlled trial design. The maintenance intervention will reinforce and extend the messages of Family Connections related to strategies to address the home environment, parenting skills to promote healthy eating and activity, and parental modeling of appropriate eating and PA. Changes in BMI percentile ranking will be used as the primary outcome. Other key outcomes will be PA and eating behaviors (i.e., compares Family Connections alone to Family Connections plus automated telephone follow-up)

SECONDARY AIM 1: Compare the effectiveness of each intervention condition to positively change parental BMI, PA, and eating behaviors. Second, by omitting the overweight child from the intervention process significant reductions in the child's reporting of eating disorder symptoms were found when compared to intervention models that included the child as a primary agent of personal change.

SECONDARY AIM 2: Determine the effectiveness of Family Connections (with and without follow-up) to decrease child eating disorder symptoms when compared to standard care

Study Measures:

Measures were collected from the child and parent at the baseline study visit; at the 6 month study visit; and at the 12 month study visit.

Child:

* height and weight
* accelerometer (measure of physical activity)
* self efficacy questions
* subjective measures of screen time and physical activity
* Kids Eating Disorders Survey (KEDS)
* Pediatric Quality of Life survey (PEDSQL)
* Block dietary recall survey

Parent:

* Height and weight
* Fat and Fibre survey
* Demographic information
* Self efficacy questions
* Health literacy questions
* Rapid Assessment of Physical Activity (RAPA)
* Home Environment survey
* Family health history
* Quality of life questions

During the 6 month assessment, parents (regardless of study arm assigned) were given a short survey to complete regarding their level of interest and satisfaction of IVR. At the 12 month assessment, parents completed a satisfaction survey regarding their experience with the study process.

ELIGIBILITY:
Inclusion Criteria:

* All boys and girls within the KPCO HMO system of the greater Denver area who are between the ages of 8 and 12 at the time of the initial assessment with a BMI of 85% or above.

Exclusion Criteria:

* Parents for whom English is not their language of communication
* Families who intend to move within the first three months of intervention
* Families who do not have access to a telephone
* Did not agree to be randomized.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220
Dates: Start 2004-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Child BMI

SECONDARY OUTCOMES:
Parent BMI
Objective measure of physical activity using child accelorometer
Kids Eating Disorder Survey (KEDS)
Peds QOL survey
SE (self efficacy)
Self resport of physical activity
Self report of sedintary activity
Children's block food frequency survey
Parent's home environment survey
Parent self efficacy
Parent demographics
Parent QOL
Parent Rapid assessment of phycial activity (parent)
Parent Fat and Fiber survey
Parent Health Literacy
Child/family medical history
Economic survey type of medical weight management services

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Estabrooks, PhD, Principal Investigator — Kaiser-Permanente of Colorado Clinical Research Unit

REFERENCES:
- [Derived] Estabrooks PA, Shoup JA, Gattshall M, Dandamudi P, Shetterly S, Xu S. Automated telephone counseling for parents of overweight children: a randomized controlled trial. Am J Prev Med. 2009 Jan;36(1):35-42. doi: 10.1016/j.amepre.2008.09.024. PMID 19095163